CLINICAL TRIAL: NCT04874532
Title: Community Paramedicine Program to Improve Diabetes Management Among Adults Experiencing Severe Hypoglycemia
Brief Title: A Study to Improve Diabetes Management Among Adults Experiencing Severe Hypoglycemia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to deliver the intervention due to program staffing.
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rozalina G. McCoy, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-006799; R03DK127010 (NIH)
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Diabetes; Hypoglycemia; Diabetes Type 1; Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Paramedic (CP) program and Education Materials (Experimental): Subjects will receive CP home visits and telephone calls for 1 month, along with printed diabetes education materials and a resource guide for contacting their diabetes care team in addition to usual care.
  Interventions: Other: Community Paramedic Program; Other: Education Material
- Usual Care and Education Materials (Active Comparator): Subjects will receive printed diabetes education materials and a resource guide for contacting their diabetes care team in addition to usual care.
  Interventions: Other: Education Material

INTERVENTIONS:
Other: Community Paramedic Program — Patients will be seen for a 1-hr in person evaluation and follow-up will be determined on an individual basis based on patient need. During each visit, CPs will perform health status and social determinants of health assessments, physical exam, medication review/counseling, and goal setting/review.
  Arms: Community Paramedic (CP) program and Education Materials
Other: Education Material — Participants will be provided with a diabetes resource card, which will provide a list of clinic and community-based diabetes resources, along with a diabetes education packet, which will include information on diabetes self-management, healthy diet, physical activity, glucose self-monitoring, and hypoglycemia.

SUMMARY:
This pilot study will assess the feasibility, preliminary efficacy, and acceptability of the Diabetes-REM (Rescue, Engagement, and Management), a comprehensive patient-centered intervention delivered by community paramedics in the community setting to improve diabetes self-management, prevent recurrent hypoglycemia, reduce diabetes distress, and improve quality of life among adults in southeast Minnesota who have experienced severe hypoglycemia.

DETAILED DESCRIPTION:
Severe hypoglycemia in the management of diabetes is associated with high morbidity, mortality, psychological distress, and impaired quality of life. Recognizing, actively engaging, and providing comprehensive care to at-risk patients to address hypoglycemia risk factors and enhance diabetes self-management skills may help reduce the frequency/severity of hypoglycemic events, alleviate diabetes distress, and improve quality of life.

This study will assess the feasibility, preliminary efficacy, and acceptability of Diabetes-REM (Rescue, Engagement, and Management) to improve diabetes self-management among adults in southeast Minnesota who have experienced severe hypoglycemia. The D-REM program is a one month long intervention delivered by community paramedics at the patient's home. Community paramedics are trained in disease prevention, management, and wellness in addition to emergency response.

Using a two-group parallel design, 150 adults will be randomly assigned to 1 month of Diabetes-REM or usual care. Both groups will receive education materials on hypoglycemia/diabetes and clinical/community resources. One group, comprised of 75 patients, will also be cared for by community paramedics at no cost to them. Study measures will include surveys (completed by participants in both arms) and an interview (completed by a subset of participants in the arm receiving community paramedic support).

Eligible individuals who decline participation in the D-REM trial will then be offered participation in a one-time interview conducted via audio technology to understand their experiences with hypoglycemia and its prevention.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older.
* Experience of level 3 hypoglycemia
* Type 1 or type 2 diabetes.
* Paneled to a Mayo Clinic or Mayo Clinic Health System practice.
* Able to provide informed consent.
* Community-dwelling in either Freeborn, Mower, Olmsted, Steele, or Wabasha county.

Identifying patients who experienced level 3 hypoglycemia:

1. Treated by Mayo Clinic Ambulance for hypoglycemia
2. Treated in Mayo Clinic ED or hospital for hypoglycemia.
3. Patients who have a diagnosis of hypoglycemia on their electronic health record problem list.
4. Patients who experienced level 3 hypoglycemia and are referred to the community paramedic service by their healthcare provider.

Exclusion Criteria:

* Under 18 years of age.
* Cognitive impairment precluding informed consent.
* Lack of conversational English skills.
* Residency in a long-term care facility.
* Enrolled in hospice.
* Enrolled in a care coordination or disease management program.
* Advanced or terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes Self-Management | Baseline, 1 month, 4 months
  Change in Diabetes Self-Management Questionnaire (DSMQ) score

SECONDARY OUTCOMES:
Self-reported hypoglycemia | Baseline, 1 month, 4 months
  Self-reported level 1 and level 2 hypoglycemia
Health-related Quality of life (EQ-5D) | Baseline, 1 month, 4 months
  Change in EQ-5D score
Diabetes distress | Baseline, 1 month, 4 months
  Change in the Diabetes Distress Scale
Glycemic control | Baseline, 4 months
  Hemoglobin A1c level
Qualitative experience with hypoglycemia and its prevention | Baseline (one-time interview only)
  Eligible individuals who decline participation in the D-REM trial will be offered participation in a one-time interview conducted via audio technology to understand their experiences with hypoglycemia and its prevention. These interviews will be qualitatively analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Rozalina G McCoy, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhagra S, Ducharme-Smith AL, Juntunen MB, Liedl CP, Golembiewski EH, Sundt WJ, Krpata TS, Lampman MA, Espinoza AL, McCoy RR. Diabetes rescue, engagement, and management (D-REM) for hypoglycemia: Clinical trial protocol of a community paramedic program to improve diabetes management among adults with severe hypoglycemia. PLoS One. 2025 Jun 9;20(6):e0322177. doi: 10.1371/journal.pone.0322177. eCollection 2025. PMID 40489473

DOCUMENTS (1):
  • Informed Consent Form (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT04874532/ICF_000.pdf